CLINICAL TRIAL: NCT04691843
Title: Role of Iron Supplementation in Neurodevelopmental Outcome of Extremely Preterm Infants - A Pilot Study
Brief Title: Iron Supplementation and Neurodevelopmental Outcome in ELGANs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Janine Yasmin Khan, Attending Neonatologist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-4092
Record Dates: First submitted 2020-12-14; First posted 2020-12-31 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Iron-deficiency
Keywords: extreme prematurity; neurodevelopmental impairment; ferritin
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard iron dose (Active Comparator): Iron supplementation of 4mg/kg/day will start when infant is on full enteral feedings of 120-150mL/kg/day and at least two weeks old. Iron dosing will be adjusted for weight at weekly intervals to maintain dosing at 4mg/kg/day.
  Interventions: Drug: Iron Sulfate
- Early, high-dose iron (Experimental): Iron supplementation will start at 3mg/kg/day when infant is on enteral feeds of 60mL/kg/day and at least one week old, then increased to 6mg/kg/day when enteral feeds are at 100mL/kg/day. Iron dosing will be adjusted to maintain ferritin level of 70-400ng/mL. At 36 weeks corrected age, iron supplementation will be adjusted to the dose routinely used for preterm infants.
  Interventions: Drug: Iron Sulfate

INTERVENTIONS:
Drug: Iron Sulfate — Early, high dose, iron supplementation
  Other Names: Ferrous Sulfate

SUMMARY:
This study explores the relationship between iron deficiency and neurological outcome of extremely premature infants. Premature birth occurs during a critical period of brain development and maturation, and before adequate transfer of iron across the placenta. Nutrition has a significant impact on ultimate outcome of survivors of prematurity. One of the biomarkers of nutrition in the premature infant is iron, and iron supplementation is essential for growth and brain development at low gestational age. As a result, the Committee on Nutrition of the American Academy of Pediatrics (AAP) recommends daily oral iron supplementation, of at least 2-4 mg/kg/day from 2 weeks of age, to prevent iron deficiency in extremely premature infants. Nevertheless, studies have shown that even with this regular care dose of iron, started from 2 weeks of age, a significant number of premature infants will still develop iron-deficiency. Our hypothesis states that starting high dose iron supplementation early will improve neurological development and outcome in extremely premature infants (those born at less than 28 weeks gestational age). This study will provide data showing whether individualized iron supplementation using higher doses of iron, started earlier (after the first week of life) when guided by periodic screening of their body's iron status with ferritin levels, will mitigate iron deficiency and promote improved neurodevelopmental outcome in this vulnerable infant population.

DETAILED DESCRIPTION:
This is a prospective, randomized, unblinded, controlled study of early, high-dose iron for neuroprotection in extremely preterm infants born between 24 0/7 weeks and 30 6/7 weeks gestation. This study has chosen to study newborns between 24-0/7 and 30-6/7 weeks of gestation because of (1) high likelihood of poor outcome, (2) highest risk of iron deficiency and potentially most likely to benefit from intervention based on their stage of brain development, (3) previously studied to assess safety of this iron regimen in Preterm Erythropoietin Neuroprotection Trial (PENUT) protocol, and (4) absence of therapeutic interventions to improve neurodevelopmental outcome. Study sample size is 90 patients; to be enrolled at Ann & Robert H Lurie Children's Hospital-Prentice Women's Hospital. We expect to evaluate 82 infants at 10-14 months and 22-26 months corrected age, our primary endpoints. There is no enrollment restriction based on race, ethnicity or gender. Enrollment is expected to take 18-24 months, with each subject with each subject participating through 24-26 months corrected age when final neurodevelopmental outcomes are assessed. Subjects will be randomized locally to regular-dose iron as recommended by AAP or early, high-dose iron. High-dose iron will continue until 36 weeks corrected age. Serial measurements of hemoglobin, reticulocyte count, reticulocyte hemoglobin equivalent and ferritin levels will be obtained, starting 2 weeks after starting iron supplementation, with final measurement obtained at 40 weeks corrected age or prior to discharge, whichever is first. Data will be abstracted regarding interval medical history from the electronic medical record. After discharge, Neonatal Intensive Care Unit (NICU) developmental follow-up will occur at 12 months and 24 months corrected age, at which time standardized neurodevelopmental assessments will be performed. The outcome measure is neurodevelopmental outcome at 10-14 months and 22-26 months of age. Our estimated sample size is based on the assumption that early high dose iron supplementation will reduce abnormal neurological outcome by 16%-29%, and taken together with an estimated 10% anticipated loss due to unrelated deaths, the total sample size was calculated at 90 infants (45 in each arm of the study).

ELIGIBILITY:
Inclusion Criteria:

* NICU inpatients between 24-0/7 and 30-6/7 weeks of gestation
* Infants older than one week of age and tolerating at least 60ml/kg/day of enteral feeds.
* Parental permission obtained prior to start of study

Exclusion Criteria:

* In extremis during consent window (as judged by primary attending provider)
* Known or suspected genetic disorder
* Unable to return for follow-up evaluation at 2 years of age

Ages: 7 Days to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome in participants | 22-26 months corrected age
  ND impairment (NDI): defined as the presence of any of the following: Bayley Scales of Development III Motor Standard Score, Language or Cognitive Standard Score < 70 (severe, 2 standard deviations (SD) below mean) or < 85 (moderate, 1 SD below mean)

SECONDARY OUTCOMES:
Iron insufficiency as assessed by ferritin level (ng/mL) | At discharge or 40 weeks corrected age (whichever occurs first), up to 16 weeks
  Iron insufficiency will be determined by ferritin level less than 70 ng/mL
Iron insufficiency as assessed by hemoglobin level (g/dL) | At discharge or 40 weeks corrected age (whichever occurs first), up to 16 weeks
  Iron insufficiency will be determined by hemoglobin level less than 8 g/dL
Iron insufficiency as assessed by reticulocyte hemoglobin equivalent (Ret-He, pg) | At discharge or 40 weeks corrected age (whichever occurs first), up to 16 weeks
  Iron insufficiency will be determined by Ret-He less than 27.2 pg
Iron insufficiency as assessed by reticulocyte count (%) | At discharge or 40 weeks corrected age (whichever occurs first), up to 16 weeks
  Iron insufficiency will be determined by reticulocyte count less than 2%

OTHER OUTCOMES:
Assess whether measurement of ferritin (ng/mL) or hemoglobin (g/dL) is superior in guiding intervention of iron-insufficiency | Throughout hospitalization, up to 16 weeks
  Assess whether measurement of ferritin (ng/mL) and adjustment of iron dosing to maintain normal ferritin level of 70-400 ng/mL, compared to measurement of hemoglobin alone, is superior in response to iron-insufficiency
Assess whether measurement of ferritin (ng/mL) or reticulocyte count (%) is superior in guiding intervention of iron-insufficiency | Throughout hospitalization, up to 16 weeks
  Assess whether measurement of ferritin (ng/mL) and adjustment of iron dosing to maintain normal ferritin level of 70-400 ng/dL, compared to measurement of reticulocyte count (%) alone, is superior in response to iron-insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Janine Y Khan, MD, MBA, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IDP available.